CLINICAL TRIAL: NCT06994013
Title: Acute Effects of High- vs. Low-frequency Vibration Foam Rolling on Flexibility, Dynamic Balance and Vertical Jump in Young Male Recreational Athletes: a Randomized Controlled Cross-over Study Design
Brief Title: Acute Effects of High- vs. Low-frequency Vibration Foam Rolling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Erhan Seçer, Principal Investigator, Celal Bayar University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: CBU-FTR-ES-O6
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Myofascial Release
Keywords: Recreational athletes; Flexibility; Dynamic balance; Vertical jump

STUDY DESIGN:
Intervention Model Description: Randomized controlled cross-over study design
Who Masked: Outcomes Assessor
Masking Description: Outcome measures assessments will be performed by an investigator who is blinded to group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HFVFR Group (Active Comparator): Athletes will be performed three sets of HFVFR for 30 s, with a 30 s break between each set and exercise. The rolling frequency will be standardized using a metronome set at 60 beats per minute. Athletes will be instructed to roll at a velocity of two metronome beats for each rolling direction. Intensity of pressure will be controlled with a target rating of 7 of 10 on a Numerical Rating Scale (0 = no discomfort and 10 = maximum discomfort) during HFVFR intervention. The target muscle groups and/or body sides will be anterior thigh, posterior thigh, posterior calf, iliotibial-band, and gluteals (buttocks).During HFVFR, the vibrator booster will be set to a frequency of 67 hz, which is within the optimal frequency range (12 to 90 hz) to influence musculoskeletal system, and an amplitude of 1.95 mm.
  Interventions: Other: High-frequency vibration foam rolling
- LFVFR Group (Active Comparator): Athletes will be performed three sets of LFVFR for 30 s, with a 30 s break between each set and exercise. The rolling frequency will be standardized using a metronome set at 60 beats per minute. Athletes will be instructed to roll at a velocity of two metronome beats for each rolling direction. Intensity of pressure will be controlled with a target rating of 7 of 10 on a Numerical Rating Scale (0 = no discomfort and 10 = maximum discomfort) during LFVFR intervention. The target muscle groups and/or body sides will be anterior thigh, posterior thigh, posterior calf, iliotibial-band, and gluteals (buttocks).During LFVFR, the vibrator booster will be set to a frequency of 35 hz, which is within the optimal frequency range (12 to 90 hz) to influence musculoskeletal system, and an amplitude of 1.95 mm.
  Interventions: Other: Low-frequency vibration foam rolling
- Control Group (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Other: High-frequency vibration foam rolling — Athletes will be performed three sets of HFVFR for 30 s, with a 30 s break between each set and exercise. The rolling frequency will be standardized using a metronome set at 60 beats per minute. Athletes will be instructed to roll at a velocity of two metronome beats for each rolling direction. Intensity of pressure will be controlled with a target rating of 7 of 10 on a Numerical Rating Scale (0 = no discomfort and 10 = maximum discomfort) during HFVFR intervention. The target muscle groups and/or body sides will be anterior thigh, posterior thigh, posterior calf, iliotibial-band, and gluteals (buttocks).During HFVFR, the vibrator booster will be set to a frequency of 67 hz, which is within the optimal frequency range (12 to 90 hz) to influence musculoskeletal system, and an amplitude of 1.95 mm.
  Arms: HFVFR Group
Other: Low-frequency vibration foam rolling — Athletes will be performed three sets of LFVFR for 30 s, with a 30 s break between each set and exercise. The rolling frequency will be standardized using a metronome set at 60 beats per minute. Athletes will be instructed to roll at a velocity of two metronome beats for each rolling direction. Intensity of pressure will be controlled with a target rating of 7 of 10 on a Numerical Rating Scale (0 = no discomfort and 10 = maximum discomfort) during LFVFR intervention. The target muscle groups and/or body sides will be anterior thigh, posterior thigh, posterior calf, iliotibial-band, and gluteals (buttocks).During LFVFR, the vibrator booster will be set to a frequency of 35 hz, which is within the optimal frequency range (12 to 90 hz) to influence musculoskeletal system, and an amplitude of 1.95 mm.
  Arms: LFVFR Group

SUMMARY:
This study aims to compare the acute effects of low- and high-frequency vibration foam rolling on flexibility, dynamic balance, and vertical jump in young male recreational athletes. Fourteen athletes will be included in this study, planned as a randomized controlled cross-over study. All athletes wil be completed three interventions: 1) low-frequency vibration foam rolling (LFVFR), 2) high-frequency vibration foam rolling (HFVFR), 3) rest control. Pre- and post-test assessment will be included flexibilty, assessed with the sit-and-reach test; dynamic balance, assessed with the Y balance test; and vertical jump, assessed with the vertical jump test.

ELIGIBILITY:
Inclusion Criteria:

* To volunteer to participate in the study
* To engage in sports activities at least 2-3 days a week

Exclusion Criteria:

* Players with a history of major sports injury or time-loss injury that required surgery
* Musculoskeletal problems that compromised their performance in the study
* A history of lower extremity pathology in the 3 months before the study
* used any drugs or supplements

Ages: 20 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Flexibility | two weeks
  Flexibility will be assessed with the sit-and-reach test using an adjustable sit-and-reach bench (Adjustable Sit-and-Reach Flexibility Tester, Lafayette Instrument Company, Lafayette IN, USA). The sit-and-reach test is a valid and reliable method used to assess flexibility in many studies. First, the sit-and-reach bench placed on the mat will be fixed to the wall, and the players will be asked to place the soles of their feet on the sit-reach bench with their knees completely straight on the mat. Then, after one trial, players will be asked to reach forward as far as possible three times without bending their knees, and the average of the three assessments will be used for analysis.

SECONDARY OUTCOMES:
Dynamic balance | two weeks
  Dynamic balance will be assessed with the Y balance test. Before the assessment, the players will be performed three trials each with 30-second rest intervals for the dominant extremity, and after the trials, the players will be given a five-minute recovery period. During the assessment after the recovery process, to ensure standardization, the players will be asked to position their dominant extremity at the centre of the junction of the measuring tapes, lie on the measuring tape with their non-dominant extremity, extending as far as possible in the anterior, posterolateral, and posteromedial directions, and touch the furthest point they could reach with their toes. This procedure will be performed by players three times with 30-second rest intervals. The greater reach distance for each direction will be calculated with the formula [(reaching distance/lower extremity length) x 100 = percentage of the maximum reaching distance)], and will be normalised with the extremity length.
Vertical jump | two weeks
  Vertical jump will be assessed with the Performanz JumpR, a valid and reliable device for assessing different jump performances.This device measures jump height based on the individual's flight time using the equation (jump height= 980.6653(flight time/1000.0)2/8). It also calculates anaerobic power using the individual's weight, flight time, and contact time using the equation (anaerobic power=weight x [9.813(flight time/2000,000)/(contact time/1000)]). For each jump, subjects will be instructed to jump as high as possible and keep their hands on their hips. There will be 1 minute of rest between jumps. All athletes will be received instructions to maximize their jump height and were verbally encouraged to exert maximum effort during all jump trials. The average of the three assessments will be used for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar University, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.